CLINICAL TRIAL: NCT07334327
Title: Efficacy of eXtracorPoreal bLOod puRification Using oXiris in Patients With SEptic Shock: A Multicenter Propensity-matched Cohort Study (EXPOLRE Study)
Brief Title: Extracorporeal Blood Purification Using Oxiris for Septic Shock (EXPLORE Study)
Acronym: EXPOLRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Collaborators: Vantive Health LLC (Industry)
Responsible Party: Principal Investigator, Woo Hyun Cho, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-2025-005
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Septic Shock; Multi Organ Failure
Keywords: Septic shock; multi organ failure; blood purification; cytokine
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: This is a multicenter, single-arm interventional study designed to evaluate the efficacy of Oxiris-based blood purification therapy in patients with septic shock. To evaluate the treatment effect, the study will use an external control group from the Korean Sepsis Alliance (KSA) registry, a large-scale prospective observational cohort. Researchers will apply 1:2 propensity score matching based on age, sex, comorbidities, initial SOFA score, and site of infection to compare the Oxiris-treated group with the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxiris Treatment Group (Experimental): Participants in this arm will receive extracorporeal blood purification therapy using the Oxiris filter (Baxter) for the management of septic shock. The intervention consists of continuous venovenous hemodiafiltration (CVVHDF) for up to 72 hours, with the Oxiris filter replaced every 24 hours to maximize adsorption efficacy. For patients not requiring renal replacement therapy (RRT), slow continuous ultrafiltration (SCUF) will be performed for adsorption therapy only. All participants will also receive standard intensive care according to institutional protocols.
  Interventions: Device: Oxiris Filter (Blood Purification Device)

INTERVENTIONS:
Device: Oxiris Filter (Blood Purification Device) — The Oxiris filter (Baxter) will be used for extracorporeal blood purification in patients with septic shock.
  * Standard Procedure: All participants will undergo continuous venovenous hemodiafiltration (CVVHDF) or slow continuous ultrafiltration (SCUF) depending on the need for renal replacement therapy (RRT).
  * Oxiris Protocol: To maximize the adsorption efficacy of endotoxins and cytokines, the Oxiris filter will be replaced every 24 hours.
  * Duration: The treatment will continue for up to 72 hours (total of 3 filters per participant).
  * Control Comparison: The outcomes of this intervention group will be compared with a propensity score-matched control group from the Korean Sepsis Alliance (KSA) registry who received standard care without Oxiris.
  Other Names: Oxiris hemofilter; AN69ST based filter

SUMMARY:
The goal of this clinical trial is to evaluate if a blood purification treatment called "Oxiris" works to help adults with septic shock. The main questions it aims to answer are: (1) Does Oxiris treatment lower the risk of death or organ failure within the first 7 days? (2) Does Oxiris treatment lower the level of inflammation in the body? Researchers will compare participants who receive Oxiris treatment to a group of participants who receive standard medical care to see if Oxiris helps them recover better.

Participants will:

1. Receive blood purification therapy using the Oxiris filter for up to 3 days while in the intensive care unit (ICU).
2. Have their blood tested at the start of the study and 3 days later to check for inflammation and organ function.
3. Be followed by the research team for about 30 days to check on their health and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 19 years of age or older.
* Participants must be diagnosed with septic shock (a severe body-wide response to infection that leads to dangerously low blood pressure).
* Participants must be in a condition where the medical team has decided that blood purification therapy (like CRRT) is necessary.

Exclusion Criteria:

* People who have a "Do Not Resuscitate" (DNR) order or are not expected to survive more than 24 hours.
* People who are pregnant or breastfeeding.
* People who are known to be allergic to the materials used in the Oxiris filter (such as heparin or specific plastics).
* People who are already participating in another clinical trial that might affect the results of this study.
* People whom the doctor decides are not suitable for the study for other medical safety reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of early organ dysfunction and mortality at Day 7 | 7 days after treatment initiation
  This is a composite outcome defined as either an increase in Sequential Organ Failure Assessment (SOFA) score of 2 points or more from baseline, or death from any cause, within 7 days after the start of Oxiris treatment. The SOFA score measures the function of six organ systems (respiratory, cardiovascular, hepatic, coagulation, renal, and neurological), with higher scores indicating more severe organ dysfunction.

SECONDARY OUTCOMES:
All-cause mortality | Day 28
  Percentage of participants who died from any cause
Change in Sequential Organ Failure Assessment(SOFA) score | Day 3
  Change in the Sequential Organ Failure Assessment (SOFA) score from baseline to Day 3 (Higher scores mean a worse outcome)
Change in Procalcitonin | Day 3
  Change in serum procalcitonin levels as an inflammatory marker
Change in IL-6 | Day 3
  Change in Interleukin-6 levels (if measured).

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect the privacy of study participants. The data contains sensitive clinical information, and the current IRB approval and informed consent do not include provisions for public data sharing with external researchers.